CLINICAL TRIAL: NCT03432663
Title: Using Time-dependent Intravenous Infusions of Amiodarone for Conversions to Sinus Rhythms in Patients With Paroxysmal Atrial Fibrillation
Brief Title: Time-dependent Amiodarone Treatment in Atrial Fibrillation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto de Cardiología y Medicina Vascular Hospital Zambrano-Hellion Tec Salud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-LS002
Record Dates: First submitted 2018-01-29; First posted 2018-02-14 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Intravenous Amiodarone; Drug safety profile; Chemical cardioversion
MeSH Terms: conditions — Atrial Fibrillation | interventions — Amiodarone

STUDY DESIGN:
Intervention Model Description: 60 emergency adult patients who were candidates for drug cardioversion after first symptomatic episodes of Atrial fibrillation to either (1)24 hour continuous infusion or (2)72 hours continuous intravenous Amiodarone or until sinus rhythms was reached.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 24h infusion (Experimental): Intravenous amiodarone infusions at doses of 5 mg/Kg for over 30 min, followed by 20 mg/Kg until 24 h was reached Intravenous amiodarone (1)
  Interventions: Drug: Intravenous amiodarone(1)
- 72h infusion (Experimental): Intravenous amiodarone infusions at doses of 5 mg/Kg for over 30 min, followed by 20 mg/Kg every 24 h for up to 72 h or until sinus rhythm was reached Intravenous amiodarone (2)
  Interventions: Drug: Intravenous amiodarone(2)

INTERVENTIONS:
Drug: Intravenous amiodarone(1) — Intravenous amiodarone infusions at doses of 5 mg/Kg for over 30 min, followed by 20 mg/Kg until 24 h was reached
  Other Names: 24 hour amiodarone
  Arms: 24h infusion
Drug: Intravenous amiodarone(2) — Intravenous amiodarone infusions at doses of 5 mg/Kg for over 30 min, followed by 20 mg/Kg every 24 h for up to 72 h or until sinus rhythm was reached
  Other Names: 72 hour amiodarone
  Arms: 72h infusion

SUMMARY:
Sixty consecutive emergency patients with newly diagnosed Atrial Fibrillation were randomized into two groups. The first received intravenous amiodarone infusions continuously for 24 hours; the second received Amiodarone until sinus rhythms was reached or for up to 72 hours.

The efficacy and safety of administering intravenous infusions of amiodarone for up to 72 hours were investigated and compared to the efficacy and safety of administering a standard 24 hours infusion of amiodarone. Specifically, the use of up to 72 hours infusions was considered as a new strategy to improve rates of conversion to sinus rhythm without altering the safety profile of the drug.

DETAILED DESCRIPTION:
An open randomized clinical trial was conducted that included 60 emergency adult patients who were candidates for drug cardioversion after first symptomatic episodes of AF.

The patients were randomized in equal proportions and sequentially placed in one of two treatment groups; no patient knew to which group he or she belonged. The first group received intravenous amiodarone infusions at doses of 5 mg/Kg for over 30 min, followed by 20 mg/Kg until 24 hours was reached. The second group received intravenous amiodarone infusions at doses of 5 mg/Kg for over 30 min, followed by 20 mg/Kg every 24 hours for up to 72 hours.

All patients were continuously monitored using electrocardiograms, and echocardiograms were performed within 24 hours after the randomized trial began. The exact time of each patient's cardioversion was documented. In addition, general laboratory tests, lipid profiles, thyroid profiles and chest X-rays were obtained for all patients.

A sample size of 30 subjects in each group was calculated. A conversion rate of 60% was assumed, according to literature, and an estimated increase to 90% was assumed for the experimental group to find differences with a power of 0.8 and an alpha error of 0.05.

The primary goal was to obtain was a sinus rhythm conversion rate. The secondary goal was to obtain a combined complication rate by noting various complications in the patients, such as phlebitis, symptomatic hypotension that required vasopressors, bradycardia, nausea, vomiting and any organ embolism.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Emergency patients
* First symptomatic episodes of Atrial Fibrillation

Exclusion Criteria:

* Hemodynamic instability,
* Previous use of antiarrhythmic drugs
* Use of digoxin seven or fewer days prior to the study
* Active thyroid disease
* Known adverse reactions to amiodarone
* Other ventricular arrhythmias
* Contraindications for anticoagulation
* Acute renal failure
* Chronic liver disease
* Transaminase levels that were twice the normal levels
* Acute pulmonary edema
* Uncontrolled hypertension (> 180/110 mmHg)
* Unstable angina
* Patients who were pregnant and/or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-08-01 (Actual); Primary Completion 2009-11-30 (Actual); Study Completion 2009-11-30 (Actual)

PRIMARY OUTCOMES:
Obtain a continuous sinus rhythm | 72 hours
  Monitoring using continuous telemetry.

SECONDARY OUTCOMES:
Complication rate of continuous amiodarone intravenous infusion | 72 hours
  Obtain a combined complication rate by noting various complications in the patients, such as phlebitis, symptomatic hypotension that required vasopressors, bradycardia, nausea, vomiting and any organ embolism.

CONTACTS AND LOCATIONS:
Overall Officials: Luis A Sanchez-Trujillo, MD, Principal Investigator — Escuela de Medicina y Ciencias de la Salud. Tecnológico de Monterrey. Monterrey. México
Locations (1):
- Hospital Universitario "Dr. José Eleuterio González". Universidad Autónoma de Nuevo León, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cotter G, Blatt A, Kaluski E, Metzkor-Cotter E, Koren M, Litinski I, Simantov R, Moshkovitz Y, Zaidenstein R, Peleg E, Vered Z, Golik A. Conversion of recent onset paroxysmal atrial fibrillation to normal sinus rhythm: the effect of no treatment and high-dose amiodarone. A randomized, placebo-controlled study. Eur Heart J. 1999 Dec;20(24):1833-42. doi: 10.1053/euhj.1999.1747. PMID 10581142
- [Background] Snow V, Weiss KB, LeFevre M, McNamara R, Bass E, Green LA, Michl K, Owens DK, Susman J, Allen DI, Mottur-Pilson C; AAFP Panel on Atrial Fibrillation; ACP Panel on Atrial Fibrillation. Management of newly detected atrial fibrillation: a clinical practice guideline from the American Academy of Family Physicians and the American College of Physicians. Ann Intern Med. 2003 Dec 16;139(12):1009-17. doi: 10.7326/0003-4819-139-12-200312160-00011. PMID 14678921
- [Background] Joseph AP, Ward MR. A prospective, randomized controlled trial comparing the efficacy and safety of sotalol, amiodarone, and digoxin for the reversion of new-onset atrial fibrillation. Ann Emerg Med. 2000 Jul;36(1):1-9. doi: 10.1067/mem.2000.107655. PMID 10874228
- [Background] Tuseth V, Jaatun HJ, Dickstein K. Amiodarone infusion in the treatment of acute atrial fibrillation or flutter: high versus low dose treatment. Heart. 2005 Jul;91(7):964-5. doi: 10.1136/hrt.2004.049171. No abstract available. PMID 15958375
- [Background] Waldo AL. Management of atrial fibrillation: the need for AFFIRMative action. AFFIRM investigators. Atrial Fibrillation Follow-up Investigation of Rhythm Management. Am J Cardiol. 1999 Sep 15;84(6):698-700. doi: 10.1016/s0002-9149(99)00419-1. No abstract available. PMID 10498142
- [Background] Wyse DG, Waldo AL, DiMarco JP, Domanski MJ, Rosenberg Y, Schron EB, Kellen JC, Greene HL, Mickel MC, Dalquist JE, Corley SD; Atrial Fibrillation Follow-up Investigation of Rhythm Management (AFFIRM) Investigators. A comparison of rate control and rhythm control in patients with atrial fibrillation. N Engl J Med. 2002 Dec 5;347(23):1825-33. doi: 10.1056/NEJMoa021328. PMID 12466506
- [Background] Go AS, Hylek EM, Phillips KA, Chang Y, Henault LE, Selby JV, Singer DE. Prevalence of diagnosed atrial fibrillation in adults: national implications for rhythm management and stroke prevention: the AnTicoagulation and Risk Factors in Atrial Fibrillation (ATRIA) Study. JAMA. 2001 May 9;285(18):2370-5. doi: 10.1001/jama.285.18.2370. PMID 11343485
- [Background] Benjamin EJ, Wolf PA, D'Agostino RB, Silbershatz H, Kannel WB, Levy D. Impact of atrial fibrillation on the risk of death: the Framingham Heart Study. Circulation. 1998 Sep 8;98(10):946-52. doi: 10.1161/01.cir.98.10.946. PMID 9737513
- [Background] Vaziri SM, Larson MG, Benjamin EJ, Levy D. Echocardiographic predictors of nonrheumatic atrial fibrillation. The Framingham Heart Study. Circulation. 1994 Feb;89(2):724-30. doi: 10.1161/01.cir.89.2.724. PMID 8313561
- [Background] Kumana CR, Cheung BM, Cheung GT, Ovedal T, Pederson B, Lauder IJ. Rhythm vs. rate control of atrial fibrillation meta-analysed by number needed to treat. Br J Clin Pharmacol. 2005 Oct;60(4):347-54. doi: 10.1111/j.1365-2125.2005.02449.x. PMID 16187966
- [Background] Lim HS, Hamaad A, Lip GY. Clinical review: clinical management of atrial fibrillation - rate control versus rhythm control. Crit Care. 2004 Aug;8(4):271-9. doi: 10.1186/cc2827. Epub 2004 Feb 19. PMID 15312210
- [Background] Chevalier P, Durand-Dubief A, Burri H, Cucherat M, Kirkorian G, Touboul P. Amiodarone versus placebo and class Ic drugs for cardioversion of recent-onset atrial fibrillation: a meta-analysis. J Am Coll Cardiol. 2003 Jan 15;41(2):255-62. doi: 10.1016/s0735-1097(02)02705-5. PMID 12535819
- [Background] Hauser TH, Pinto DS, Josephson ME, Zimetbaum P. Early recurrence of arrhythmia in patients taking amiodarone or class 1C agents for treatment of atrial fibrillation or atrial flutter. Am J Cardiol. 2004 May 1;93(9):1173-6. doi: 10.1016/j.amjcard.2004.01.051. PMID 15110217
- [Background] Khan IA, Mehta NJ, Gowda RM. Amiodarone for pharmacological cardioversion of recent-onset atrial fibrillation. Int J Cardiol. 2003 Jun;89(2-3):239-48. doi: 10.1016/s0167-5273(02)00477-1. PMID 12767548
- [Background] Hagens VE, Van Gelder IC, Crijns HJ; RAte Control Versus Electrical Cardioversion Of Persistent Atrial Fibrillation (RACE) Study Group. The RACE study in perspective of randomized studies on management of persistent atrial fibrillation. Card Electrophysiol Rev. 2003 Jun;7(2):118-21. doi: 10.1023/a:1027439430017. PMID 14618033
- [Background] McNamara RL, Tamariz LJ, Segal JB, Bass EB. Management of atrial fibrillation: review of the evidence for the role of pharmacologic therapy, electrical cardioversion, and echocardiography. Ann Intern Med. 2003 Dec 16;139(12):1018-33. doi: 10.7326/0003-4819-139-12-200312160-00012. PMID 14678922
- [Background] Maisel WH, Kuntz KM, Reimold SC, Lee TH, Antman EM, Friedman PL, Stevenson WG. Risk of initiating antiarrhythmic drug therapy for atrial fibrillation in patients admitted to a university hospital. Ann Intern Med. 1997 Aug 15;127(4):281-4. doi: 10.7326/0003-4819-127-4-199708150-00004. PMID 9265427
- [Background] Kreiss Y, Sidi Y, Gur H. Efficacy and safety of intravenous amiodarone in recent-onset atrial fibrillation: experience in patients admitted to a general internal medicine department. Postgrad Med J. 1999 May;75(883):278-81. doi: 10.1136/pgmj.75.883.278. PMID 10533631
- [Background] Xanthos T, Bassiakou E, Vlachos IS, Bassiakos S, Michalakis K, Moutzouris DA, Papadimitriou L. Intravenous and oral administration of amiodarone for the treatment of recent onset atrial fibrillation after digoxin administration. Int J Cardiol. 2007 Oct 18;121(3):291-5. doi: 10.1016/j.ijcard.2007.02.024. Epub 2007 Apr 16. PMID 17434635
- [Background] Vardas PE, Kochiadakis GE, Igoumenidis NE, Tsatsakis AM, Simantirakis EN, Chlouverakis GI. Amiodarone as a first-choice drug for restoring sinus rhythm in patients with atrial fibrillation: a randomized, controlled study. Chest. 2000 Jun;117(6):1538-45. doi: 10.1378/chest.117.6.1538. PMID 10858380
- [Background] Hohnloser SH, Kuck KH, Lilienthal J. Rhythm or rate control in atrial fibrillation--Pharmacological Intervention in Atrial Fibrillation (PIAF): a randomised trial. Lancet. 2000 Nov 25;356(9244):1789-94. doi: 10.1016/s0140-6736(00)03230-x. PMID 11117910
- [Background] Bernard EO, Schmid ER, Schmidlin D, Scharf C, Candinas R, Germann R. Ibutilide versus amiodarone in atrial fibrillation: a double-blinded, randomized study. Crit Care Med. 2003 Apr;31(4):1031-4. doi: 10.1097/01.CCM.0000053555.78624.0F. PMID 12682468
- [Background] Thomas SP, Guy D, Wallace E, Crampton R, Kijvanit P, Eipper V, Ross DL, Cooper MJ. Rapid loading of sotalol or amiodarone for management of recent onset symptomatic atrial fibrillation: a randomized, digoxin-controlled trial. Am Heart J. 2004 Jan;147(1):E3. doi: 10.1016/s0002-8703(03)00526-x. PMID 14691441
- [Background] Decker WW, Smars PA, Vaidyanathan L, Goyal DG, Boie ET, Stead LG, Packer DL, Meloy TD, Boggust AJ, Haro LH, Laudon DA, Lobl JK, Sadosty AT, Schears RM, Schiebel NE, Hodge DO, Shen WK. A prospective, randomized trial of an emergency department observation unit for acute onset atrial fibrillation. Ann Emerg Med. 2008 Oct;52(4):322-8. doi: 10.1016/j.annemergmed.2007.12.015. Epub 2008 Mar 14. PMID 18339449
- [Background] del Arco C, Martin A, Laguna P, Gargantilla P; Investigators in the Spanish Atrial Fibrillation in Emergency Medicine Study Group (GEFAUR). Analysis of current management of atrial fibrillation in the acute setting: GEFAUR-1 study. Ann Emerg Med. 2005 Nov;46(5):424-30. doi: 10.1016/j.annemergmed.2005.03.002. Epub 2005 May 31. PMID 16271674
- [Background] Carlsson J, Miketic S, Windeler J, Cuneo A, Haun S, Micus S, Walter S, Tebbe U; STAF Investigators. Randomized trial of rate-control versus rhythm-control in persistent atrial fibrillation: the Strategies of Treatment of Atrial Fibrillation (STAF) study. J Am Coll Cardiol. 2003 May 21;41(10):1690-6. doi: 10.1016/s0735-1097(03)00332-2. PMID 12767648
- [Background] Roy D, Talajic M, Nattel S, Wyse DG, Dorian P, Lee KL, Bourassa MG, Arnold JM, Buxton AE, Camm AJ, Connolly SJ, Dubuc M, Ducharme A, Guerra PG, Hohnloser SH, Lambert J, Le Heuzey JY, O'Hara G, Pedersen OD, Rouleau JL, Singh BN, Stevenson LW, Stevenson WG, Thibault B, Waldo AL; Atrial Fibrillation and Congestive Heart Failure Investigators. Rhythm control versus rate control for atrial fibrillation and heart failure. N Engl J Med. 2008 Jun 19;358(25):2667-77. doi: 10.1056/NEJMoa0708789. PMID 18565859
- [Background] Galve E, Rius T, Ballester R, Artaza MA, Arnau JM, Garcia-Dorado D, Soler-Soler J. Intravenous amiodarone in treatment of recent-onset atrial fibrillation: results of a randomized, controlled study. J Am Coll Cardiol. 1996 Apr;27(5):1079-82. doi: 10.1016/0735-1097(95)00595-1. PMID 8609324
- [Background] Wolf PA, Abbott RD, Kannel WB. Atrial fibrillation as an independent risk factor for stroke: the Framingham Study. Stroke. 1991 Aug;22(8):983-8. doi: 10.1161/01.str.22.8.983. PMID 1866765
- [Background] Martinez-Marcos FJ, Garcia-Garmendia JL, Ortega-Carpio A, Fernandez-Gomez JM, Santos JM, Camacho C. Comparison of intravenous flecainide, propafenone, and amiodarone for conversion of acute atrial fibrillation to sinus rhythm. Am J Cardiol. 2000 Nov 1;86(9):950-3. doi: 10.1016/s0002-9149(00)01128-0. PMID 11053705
- [Background] Kochiadakis GE, Igoumenidis NE, Hamilos ME, Marketou ME, Chlouverakis GI, Vardas PE. A comparative study of the efficacy and safety of procainamide versus propafenone versus amiodarone for the conversion of recent-onset atrial fibrillation. Am J Cardiol. 2007 Jun 15;99(12):1721-5. doi: 10.1016/j.amjcard.2007.01.059. Epub 2007 Apr 26. PMID 17560882
- [Background] Cybulski J, Kulakowski P, Budaj A, Danielewicz H, Maciejewicz J, Kawka-Urbanek T, Ceremuzynski L. Intravenous amiodarone for cardioversion of recent-onset atrial fibrillation. Clin Cardiol. 2003 Jul;26(7):329-35. doi: 10.1002/clc.4950260707. PMID 12862299
- [Background] Hilleman DE, Spinler SA. Conversion of recent-onset atrial fibrillation with intravenous amiodarone: a meta-analysis of randomized controlled trials. Pharmacotherapy. 2002 Jan;22(1):66-74. doi: 10.1592/phco.22.1.66.33492. PMID 11794432
- [Background] National Clinical Guideline Centre (UK). Atrial Fibrillation: The Management of Atrial Fibrillation. London: National Institute for Health and Care Excellence (UK); 2014 Jun. Available from http://www.ncbi.nlm.nih.gov/books/NBK248059/ PMID 25340239
- [Background] January CT, Wann LS, Alpert JS, Calkins H, Cigarroa JE, Cleveland JC Jr, Conti JB, Ellinor PT, Ezekowitz MD, Field ME, Murray KT, Sacco RL, Stevenson WG, Tchou PJ, Tracy CM, Yancy CW; ACC/AHA Task Force Members. 2014 AHA/ACC/HRS guideline for the management of patients with atrial fibrillation: a report of the American College of Cardiology/American Heart Association Task Force on practice guidelines and the Heart Rhythm Society. Circulation. 2014 Dec 2;130(23):e199-267. doi: 10.1161/CIR.0000000000000041. Epub 2014 Mar 28. No abstract available. PMID 24682347
- [Background] Freemantle N, Lafuente-Lafuente C, Mitchell S, Eckert L, Reynolds M. Mixed treatment comparison of dronedarone, amiodarone, sotalol, flecainide, and propafenone, for the management of atrial fibrillation. Europace. 2011 Mar;13(3):329-45. doi: 10.1093/europace/euq450. Epub 2011 Jan 11. PMID 21227948
- [Background] Nadarasa K, Williams MJ. Single high oral dose amiodarone for cardioversion of recent onset atrial fibrillation. Heart Lung Circ. 2012 Aug;21(8):444-8. doi: 10.1016/j.hlc.2012.03.015. Epub 2012 May 2. PMID 22554874
- [Background] Patel DA, Lavie CJ, Milani RV, Shah S, Gilliland Y. Clinical implications of left atrial enlargement: a review. Ochsner J. 2009 Winter;9(4):191-6. PMID 21603443
- [Background] Danias PG, Caulfield TA, Weigner MJ, Silverman DI, Manning WJ. Likelihood of spontaneous conversion of atrial fibrillation to sinus rhythm. J Am Coll Cardiol. 1998 Mar 1;31(3):588-92. doi: 10.1016/s0735-1097(97)00534-2. PMID 9502640
- [Background] Emren SV, Kocabas U, Duygu H, Levent F, Simsek EC, Yapan Emren Z, Tuluce S. The role of HATCH score in predicting the success rate of sinus rhythm following electrical cardioversion of atrial fibrillation. Kardiol Pol. 2016;74(9):978-84. doi: 10.5603/KP.a2016.0044. Epub 2016 Apr 4. PMID 27040017
- [Background] Suenari K, Chao TF, Liu CJ, Kihara Y, Chen TJ, Chen SA. Usefulness of HATCH score in the prediction of new-onset atrial fibrillation for Asians. Medicine (Baltimore). 2017 Jan;96(1):e5597. doi: 10.1097/MD.0000000000005597. PMID 28072697
- [Background] Fuster V, Ryden LE, Cannom DS, Crijns HJ, Curtis AB, Ellenbogen KA, Halperin JL, Le Heuzey JY, Kay GN, Lowe JE, Olsson SB, Prystowsky EN, Tamargo JL, Wann S, Smith SC Jr, Jacobs AK, Adams CD, Anderson JL, Antman EM, Halperin JL, Hunt SA, Nishimura R, Ornato JP, Page RL, Riegel B, Priori SG, Blanc JJ, Budaj A, Camm AJ, Dean V, Deckers JW, Despres C, Dickstein K, Lekakis J, McGregor K, Metra M, Morais J, Osterspey A, Tamargo JL, Zamorano JL; American College of Cardiology; American Heart Association Task Force; European Society of Cardiology Committee for Practice Guidelines; European Heart Rhythm Association; Heart Rhythm Society. ACC/AHA/ESC 2006 guidelines for the management of patients with atrial fibrillation: full text: a report of the American College of Cardiology/American Heart Association Task Force on practice guidelines and the European Society of Cardiology Committee for Practice Guidelines (Writing Committee to Revise the 2001 guidelines for the management of patients with atrial fibrillation) developed in collaboration with the European Heart Rhythm Association and the Heart Rhythm Society. Europace. 2006 Sep;8(9):651-745. doi: 10.1093/europace/eul097. No abstract available. PMID 16987906